CLINICAL TRIAL: NCT01480817
Title: An Open Label, Phase 2 Trial Comparing Sorafenib And TACE in Advanced Hepatocellular Carcinoma With Portal Vein Invasion
Brief Title: Sorafenib VS TACE in HCC Patients With Portal Vein Invasion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty of participant enrollment.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAP
Record Dates: First submitted 2011-11-20; First posted 2011-11-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2013-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib (Active Comparator): Sorafenib 400mg po bid
  Interventions: Drug: Sorafenib
- TACE for HCC with portal vein invasion (Experimental): Antineoplastic agents are directly injected into the hepatic artery, allowing high intratumoral concentrations of drugs and thereby reducing systemic side effects. The mixture of chemotherapeutic agents and iodized oil is almost completely retained in neoplastic nodules and can remain in HCC tissue for a long time. Subsequent mechanical embolization of the artery feeding the neoplasm causes ischemic damage to the tumor and prolongs the duration of the effects of chemotherapeutic agents.
  Interventions: Procedure: TACE for HCC with portal vein invasion

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400mg po bid
  Other Names: Nexavar
  Arms: Sorafenib
Procedure: TACE for HCC with portal vein invasion — The volume of iodized oil ranged from 2 to 12 mL, and the amount of doxorubicin ranged from 10 to 60 mg. Gelatin sponge particles were mixed with mitomycin and contrast material.Cisplatin was infused at the tumor feeder vessels as a solution with a concentration of 0.5 mg/mL at a rate of 5-10 mL/min. The total amount of cisplatin used ranged from 50 to 100 mg depending on the patient's body weight and the level of infusion.
  Other Names: TACE
  Arms: TACE for HCC with portal vein invasion

SUMMARY:
The investigators are going to compare the therapeutic effect of sorafenib and transarterial chemoembolization in advanced hepatocellular carcinoma with major branch of portal vein invasion.

DETAILED DESCRIPTION:
TACE is an established therapy for patients with unresectable hepatocellular carcinoma (HCC) and has been shown to significantly improve survival in these patients compared to no treatment. Moreover, TACE can be performed safely and may improve the overall survival of patients with HCC and major branch of portal vein invasion. Sorafenib, already approved for HCC, could lead to significantly improvement in tumor control and survival in patients with advanced stage HCC. So far there are no head to head comparison reports about the efficacy of Sorafenib and TACE. Here the investigators evaluate the efficacy of sorafenib and TACE in advanced HCC with major branch of portal vein invasion.

ELIGIBILITY:
Inclusion Criteria:

1. 80 > Age >= 18 years.
2. Child-Pugh class A (class B could be included when Childs score is 7).
3. Hepatocellular carcinoma with major branch of portal vein invasion on dynamic CT or MRI

   * not only newly diagnosed treatment-naive patients,
   * but also HCC patients previously treated with other therapies in case of development of major branch of portal vein invasion
4. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements:

   * White blood cell counts (WBC) >= 2,000 /μl, Absolute neutrophil count (ANC) > 1,200/μl
   * Hemoglobin >= 8.0 g/dl
   * Platelet count > 50,000/μl
   * Serum creatinine < 1.7 mg/dl
   * Total bilirubin =< 3.0 mg/dl
   * Prothrombin Time (PT)-international normalized ratio (INR) =< 2.3 or Prothrombin Time (PT)-sec =< 6 sec
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.

Exclusion Criteria:

1. Child-Pugh score >= 8.
2. Age < 18 or >= 80 years.
3. ECOG Performance Status >= 3.
4. Recipient of living donor or deceased donor liver transplantation
5. Patients unable to understand the contents of informed consent or refuse to sign the informed consent.
6. Patients with evidence of uncontrolled or severe medical conditions requiring treatment.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to Progression (Efficacy) | every 6 weeks up to 3 years

SECONDARY OUTCOMES:
overall survival | every 6 weeks up to 3 years
objective tumor response rate | every 6 weeks up to 3 years
  Determined by dynamic-perfusion CT scan at the end of each cycle
objective tumor control rate | every 6 weeks up to 3 years
  Determined by dynamic-perfusion CT scan at the end of each cycle
progression-free survival | every 6 weeks up to 3 years
the adverse event rate and examine the toxicities | every 6 weeks up to 3 years
  The investigators will evaluate the adverse event according to Common Toxicity Criteria(version 4.0)by National Cancer Institute of National Institutes of Health
Change of perfusion parameter | every 6 weeks up to 3 years
Alpha feto protein (AFP) responsiveness | every 6 weeks up to 3 years
  AFP responder : 20% reduction from baseline AFP level after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hwan Yoon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea